CLINICAL TRIAL: NCT03941899
Title: The Analgesic Effect of Qudratus Lomborum Block II Type After Robotic-Assisted Laparoscopic Radical Prostatectomy.
Brief Title: The Analgesic Effect of QLB II After Robotic Prostatectomy. (QLB II: Quadratus Lomborum Block II Type)
Acronym: QLBII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Principal Investigator, San Salvatore Hospital of L'Aquila
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0081052
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain
Keywords: Pain, radical prostatectomy, QLB II type
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Levobupivacaine

STUDY DESIGN:
Intervention Model Description: Simon's Two-Stage single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- QLB II (Other): Quadratus Lomborum Blocck II type will be performed before robot-assisted laparoscopic radical prostatectomy
  Interventions: Other: Levobupivacaine in QLB II

INTERVENTIONS:
Other: Levobupivacaine in QLB II — Quadratus Lomborum Block II type will be performed by injecting levobupivacaine 0.375% 20 ml between latissimus dorsi and quadratus lomborum muscle.
  Other Names: Quadratus Lomborum Block II type

SUMMARY:
The analgesic effects of Quadratus Lomborum Block II type after robotic-assisted laparoscopic radical prostatectomy, will be assessed.

DETAILED DESCRIPTION:
Quadratus Lomborum Block II type will be performed before performing robotic-assisted laparoscopic radical prostatectomy.

The post-operative analgesic effect will be assessed, by using Numeric Rate Scale for pain.

The pain assessment will be evaluated during the first 24 hours from surgery. The opioids requirement and side effects will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist status I-III
* Written informed consent

Exclusion Criteria:

* Body mass Index > 35 kg/m2
* Allergies to local anesthetics
* primaries or secondaries coagulopathies
* addiction to drugs
* severe kidney and liver diseases
* cognitive impairment

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients undergoing to robotic-assisted laparoscopic radical prostatectomy
Enrollment: 48 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Analgesia | The first 24 hours from surgery
  Pain assessment by using Numeric Rate Scale for pain

SECONDARY OUTCOMES:
Opioids | The first 24 hours from surgery
  The opioids requirement (mg of equianalgesic morphine) will be assessed
Postoperative Nausea and Vomiting | The first 24 hours from surgery
  The postoperative nausea and vomiting will be assessed
Bowel function | The first 24 hours from surgery
  The recovery of bowel function will be assessed
Length of stay | Day after surgery
  The length of stay after surgery will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Franco Marinangeli, MD, Study Chair — San Salvatore Academic Hospital
Locations (1):
- San Salvatore Academic Hospital, Coppito, L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No